CLINICAL TRIAL: NCT03407989
Title: SWIDINEP a Swiss Diabetic Nephropathy Cohort
Acronym: SWIDINEP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Anne Zanchi, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CER 43/12
Record Dates: First submitted 2018-01-09; First posted 2018-01-23 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, and fresh urine samples as well as whole blood (buffy coat for DNA extraction and genotyping) are stored at -80°C in a local biobank according to the latest guidelines of the Académie Suisse des Sciences Médicales (ASSM).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With our SWIDINEP cohort, we propose to explore the relationship between vascular risk markers and renal function decline in CKD stage 1-5. In order to realize these goals, we intend to recruit 200 patients within a 7y recruitment period (2014-2021). Recruitment is done in the nephrology and diabetes ambulatory clinics in the CHUV at Lausanne. Each eligible patient is identified and whether he/she can be proposed the study is discussed with the physician in charge of the patient. Once the patient is informed and has signed the consent form, he/she is examined in the Service of Nephrology at baseline, 2y and 5y.

DETAILED DESCRIPTION:
Serum, plasma, and fresh urine samples as well as whole blood (buffy coat for DNA extraction and genotyping) are stored at -80°C in a local biobank according to the latest guidelines of the Académie Suisse des Sciences Médicales (ASSM).

The vascular phenotype includes:

* 24h ABPM with the examination of diurnal variations of blood pressure, pulse pressure and heart rate. Central pulse pressure is also calculated based on the pulse wave analysis providing information on stroke volume, central BP, aortic stiffness and arterial wave reflection. It increases with age and could expose glomerular capillaries to damage. It has been independently related to proteinuria.
* Arterial stiffness is assessed non-invasively with the commercially available Sphygmocor system (Version 8.0, At Cor Medical, Sydney, Australia) using applanation tonometry to measure carotid-femoral pulse wave velocity (PWV) and carotid and radial augmentation indexes. Pulse wave velocity is a strong surrogate for carotid-femoral arterial stiffness. Generally around 3-4m/s in the young population it increases with age. A high PWV brings to a greater transmission of pulsating pressure to the renal microcirculation and is associated with accelerated eGFR decline. Recently, a study has described its independent relationship with cardio-vascular mortality in CKD stage 2-4. Patients with a PWV at least at 10m/s had a HR for mortality of 5. Carotid and radial augmentation indexes measure the difference between the second and first systolic peak of the aortic wave and is expressed as a percentage of pulse pressure. They increase with age and have been correlated with eGFR and albuminuria.
* Carotid ultrasound is performed to assess carotid intima-media thickness. Carotid-intima media thickness is a direct measurement of atherosclerosis and can help stratify patients at CV risk. It has been associated with eGFR decline.
* Participants undergo a renal ultrasound including renal resistance index measurements as marker of intrarenal vascular disease according to a pre-specified protocol used previously in other local cohorts by the same experienced operator (PD Dr Menno Pruijm). The assessment of the intrarenal vessels is made by duplex Doppler sonography on 3 segmental arteries (superior, middle, and inferior) in each kidney. The values are then averaged to obtain the mean value for each participant. Renal resistive index (RRI) is calculated as [(peak-systolic velocity - end-diastolic velocity)/peak-systolic velocity]. The Service of nephrology has performed an important study providing reference values in a population with normal renal ultrasounds. Renal resistive index has been associated with eGFR decline. Besides, all participants are screened for underlying renal artery stenosis based on well established intrarenal Doppler criteria. The presence of other renal structural abnormalities (renal cysts, tumors, calcifications and/or hydronephrosis) is also assessed. Finally, the bladder area is systematically visualized, as well as the prostatic gland in men.
* Subjects undergo ocular examination, including best-corrected visual acuity (BCVA), slit lamp biomicroscopic exam, measurement of intraocular pressure with a non-contact tonometer and fundus examination. Choroidal thickness is measured by the EDI-OCT technique. The subfoveal choroidal thickness is measured at macular fovea from the outer portion of the hyperreflective line corresponding to the RPE to the hyporeflective line or margin corresponding to the sclerochoroidal interface. Central macular retinal thickness is determined automatically in all eyes. There are emerging data regarding the relationship of choroidal circulation and various systemic and ocular diseases. The choroid is highly vascularized tissue that supplies blood to the outer retina, including the retinal pigment epithelium (RPE) cells and photoreceptors, especially in the foveal region where there is no retinal vasculature. The choroid plays a crucial part in the physiopathology of many retinal diseases. Details of the choroidal circulation remained largely unknown due to poor resolution and reproducibility of previous choroidal imaging techniques. Imaging of the choroid was dramatically improved with the development of spectral domain optical coherence tomography and was further augmented with the advent of enhanced depth imaging. The relation between renal dysfunction and impaired ocular microcirculation remains unclear, especially in early-stage diabetes. It's been reported that the blood flow in the retinal arterioles is decreased in patients with type 2 diabetes with chronic kidney disease. Though, data on the relationship between choroidal thickness and diabetic nephropathy are sparse. As far as we are aware today, there is only one study that evaluated choroidal thickness alterations in diabetic nephropathy patients with early or no diabetic retinopathy. More precisely the subfoveal, temporal and nasal choroidal thickness was noted to be thinner in patients with diabetic nephropathy patients compared with non- diabetic nephropathy patients and normal subjects.

Quality of life questionnaires: A number of studies have shown that as kidney function decreases, disease burden increases, with lower health-related quality of life (HRQoL) for patients with late stages of chronic kidney disease. However, few studies have looked into HRQoL and its determinants in the specific population of diabetic patients with kidney disease. Assessing HRQoL and its determinants is important in chronic care as studies have shown that patients with higher HRQoL function better within the healthcare system and perform more health-promoting activities. HRQoL is assessed at baseline in patients enrolled in the cohort. The impact of baseline HRQoL on renal function decline will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* eGFR <60ml/min or albumine/creatinine ratio >3mg/mmol
* Can understand french and has signed the consent form.

Exclusion Criteria:

* Age < 18y
* Another cause of nephropathy (excluding hypertensive nephropathy, obese related nephropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with type 2 diabetes and CKD stage 1-5
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
estimated GFR decline ml/min/y | 2-5 years
  estimated GFR will be based on the creatinine based CKD-EPI formula

SECONDARY OUTCOMES:
24 hour blood pressure measurements (mmHg) and eGFR decline (ml/min/y) | 2-5 years
  Relationship of 24h blood pressure diurnal pattern and eGFR decline
Vascular markers (Pulse wave velocity (m/s); Carotid and radial augmentation indexes (%); intima media thickness (mm)) and eGFR decline (ml/min/y) | 2-5 years
  Relationship of baseline vascular markers and eGFR decline
Kidney volume (cm3) and resistance index and eGFR decline (ml/min/y) | 2-5y
  Relationship of renal volume/resistance index and eGFR decline
Biochemical parameters and eGFR decline (ml/min/y) | 2-5y
  Relationship of baseline biochemical biomarkers and eGFR decline
Genetic markers and eGFR decline (ml/min/y) | 2-5y
  Relationship of genetic markers and eGFR decline
Choroidal thickness (microm) and eGFR decline (ml/min/y) | 2-5y
  Relationship of baseline choroidal thickness and eGFR decline
Generic health-related quality of life baseline measures, CKD stage, and eGFR decline. | 2-5y
  The influence of CKD stage and eGFR decline on generic and diabetes-specific health related quality of life questionnaires.
Diabetes-specific health-related quality of life baseline measures, CKD stage, and eGFR decline. | 2-5y
  The influence of CKD stage and eGFR decline on generic and diabetes-specific health related quality of life questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland